CLINICAL TRIAL: NCT00516685
Title: A Phase II/III Trial to Assess the Safety, Immunogenicity and Preliminary Efficacy of Recombinant Human EGF-rP64K/Montanide ISA 51 Vaccine Administered to Patients With Non-Small-Cell Lung Cancer (NSCLC) After Receiving Conventional First Line Chemotherapy
Brief Title: Vaccine Therapy in Treating Patients With Non-Small Cell Lung Cancer (NSCLC) Stages IIIB/IV
Acronym: NSCLC
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Due to inability of patient enrollment, decision taken to terminate in the interests of patients and later Malaysia is incorporated into global Phase 3 trial.
Sponsor: Bioven Sdn. Bhd. (Industry)
Responsible Party: DR G SELVARATNAM, NILAI CANCER INSTITUTE
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CT 07-03
Record Dates: First submitted 2007-08-14; First posted 2007-08-15 (Estimated); Last update posted 2011-09-30 (Estimated); Status verified 2011-09

CONDITIONS: Non-small-cell Lung Cancer (NSCLC) Stage IIIb/IV
Keywords: LUNG CANCER; NSCLC; EGF; CANCER VACCINE; IMMUNOTHERAPY
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms

ARMS (2):
- Vaccine Group (Experimental): Patients in this arm will receive a low dose of Cyclophosphamide and the recombinant human rEGF-P64K/Montanide ISA 51 vaccine in addition to Best Supportive Care.
  Interventions: Biological: Recombinant Human rEGF-P64K/Montanide Vaccine
- Control Group (No Intervention): Patients in this arm will only receive Best Supportive Care.

INTERVENTIONS:
Biological: Recombinant Human rEGF-P64K/Montanide Vaccine
  Arms: Vaccine Group

SUMMARY:
The purpose of this study is to determine whether the recombinant human EGF-rP64K/Montanide ISA 51 vaccine is safe, immunogenic and effective in the treatment of stage IIIb/IV non-small-cell lung cancer (NSCLC).

ELIGIBILITY:
Inclusion Criteria:

* Patients who have signed the informed consent form.
* Patients who are eighteen years of age or over with histologically or cytologically confirmed NSCLC in advanced stages IIIb or IV, not amenable to any attempt of curative chemo-radiotherapy and/or surgery.
* Patients with measurable lesions, defined as those measurable at least in one dimension (refered to higher diameter) and with a diameter equal or higher 20 mm using conventional techniques (PET, CT scan, MRI, Rx) or equal or higher 10 mm using CT scan.
* Patients who have finished their last cycle of chemotherapy and/or radiotherapy not less than 4 weeks prior to randomization and not more than 8 weeks.
* Female patients of reproductive potential must have negative pregnancy tests. Those female volunteers admitted to the study must be using a reliable means of contraception such as tubal ligation, oral contraceptive or IUD.
* ECOG status 0 to 2.
* Patients with normal organ and bone marrow function, as defined by the parameters in accordance to that provided by the normal lab reference range.
* Patients with no evidence of objective disease progression, 1 month after finishing first line chemotherapy as per RECIST.

Exclusion Criteria:

* Patients who are candidates for combined modality treatment.
* Patients who are receiving immunosuppressive therapy including corticosteroids.
* Patients who have received immunotherapy within the previous 3 months.
* Patients who have participated in a clinical study within the previous 30 days.
* Patients who may be allergic to any component of the vaccine.
* Medical reasons considered by the investigators as disqualification from the study such as significant uncontrolled co-morbid disease or potential non-compliance with the protocol.
* Patients bearing brain metastasis from the primary lung tumor.
* Patients bearing a second primary tumor.
* Patients showing progressive disease after finishing first line chemotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2007-07

PRIMARY OUTCOMES:
Survival | Two and a half years

SECONDARY OUTCOMES:
Assessment of immunogenecity, safety as well as preliminary assessment of objective response, time of progression and quality of life | Two and a half years

CONTACTS AND LOCATIONS:
Overall Officials: G SELVARATNAM, MD, Principal Investigator — NILAI CANCER INSTITUTE
Locations (8):
- Malaysia (8):
  - Local Institution, Kubang Kerian, Kelantan
  - Local Institution, Kampung Baharu Nilai, Negeri Sembilan
  - Local Institution, Kuantan, Pahang
  - Local Institution, George Town, Pulau Pinang
  - Local Institution, Kota Kinabalu, Sabah
  - Local Institution, Klang, Selangor
  - Local Institution, Petaling Jaya, Selangor
  - Local Institution, Kuala Lumpur